CLINICAL TRIAL: NCT05567679
Title: IIT2021-09-Posadas-NA-TAZ: A Study of Tazemetostat (Tazverik) Before Prostatectomy in Men With Prostate Cancer
Brief Title: A Study of Tazemetostat (Tazverik) Before Prostatectomy in Men With Prostate Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI voluntarily closed the study.
Sponsor: Edwin Posadas, MD (Other)
Collaborators: Epizyme, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Edwin Posadas, MD, Co-Director, Experimental Therapeutics Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-09-Posadas-NA-TAZ
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Radical prostatectomy; RP
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tazemetostat (Experimental): Tazemetostat 200 mg oral tablets; 800 mg by mouth twice daily for 28 days
  Interventions: Drug: Tazverik

INTERVENTIONS:
Drug: Tazverik — Tazemetostat (Tazverik) 200 mg oral tablets; 800 mg by mouth twice daily for 28 days

SUMMARY:
This study is an open-label, single-arm, pilot, perioperative study of EZH2 inhibition in patients undergoing Radical Prostatectomy (RP). The EZH2 inhibition is intended to increase the sensitivity of the underlying tumor to the patient's immune system.

Given the absence of data in this setting, we propose to pilot this experience with 4 weeks of tazemetostat at doses known to be clinically safe and effective at inducing clinical effects via inhibition of EZH2 as established for follicular lymphoma and epithelioid sarcoma: 800 mg twice daily with or without food.

Prior to tazemetostat, blood will be collected (4 tubes) for immune cells, Circulating Tumor Cells, and plasma. This will be repeated at the time of RP. RP tissues will be collected.

Additionally, patients will have a week lead-in to wear a FitBit Charge 5TM device (or similar model) to continuously monitor physical activity from baseline up until end of study. The start of the week lead-in will be considered the baseline visit. Subjects will also be asked to continue wearing the device until end of study and option to continue for up to 2 years after end of study in follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men electing to undergo radical prostatectomy with preoperative tissue available
* Able to take oral medications
* Age ≥18 years
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate organ function
* Men with partners of childbearing potential, must have had a successful vasectomy (with medically confirmed lack of sperm that are alive) OR must either practice complete abstinence or agree to use adequate contraception
* Inclusion criteria for remote monitoring component of study with Fitbit only (failure to meet inclusion criterion for Fitbit-monitoring portion of study should not preclude participating in treatment trial): Access to a device (e.g., smart phone, tablet) that has the capability to sync to the Fitbit. Note: access can be via family member, friend, caregiver, or study-designated device provided by study member

Exclusion Criteria:

* Active intercurrent illness or malignancy requiring therapy outside of prostate cancer
* History of bleeding disorders
* Concurrent use of anti-platelet agents or therapeutic anticoagulants with the exception of low-dose aspirin (81 mg daily) or NSAIDs for pain/inflammation.

Concurrent use of strong and moderate CYP3A inhibitors and inducers

* Subjects who have previously received tazemetostat
* Currently participating in a study using an investigational, medicinal anti-cancer agent within 4 weeks prior to first dose of tazemetostat
* Exclusion criteria for remote monitoring component of study with Fitbit only (failure to meet exclusion criterion for Fitbit-monitoring portion of study should not preclude participating in treatment trial): Using a pacemaker, implantable cardiac defibrillator, neurostimulator, cochlear implants (removable hearing aids permitted), or other electronic medical equipment, per PI's discretion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, serious adverse events, and treatment-related adverse events. | From start of study treatment until confirmation of disease progression, intolerable toxicities, or withdrawal of consent, whichever came first. Assessed up to 30 days following last dose of study treatment.
  Evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Proportion of patients able to undergo surgery | At time of surgery
Proportion of patients with Grade 3 or above treatment related adverse events | From start of study treatment until confirmation of disease progression, intolerable toxicities, or withdrawal of consent, whichever came first. Assessed up to 30 days following last dose of study treatment.
  Grade 3 or above treatment related adverse events as assessed per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Proportion of patients with evaluable tissue specimens following tazemetostat | At time of surgery

SECONDARY OUTCOMES:
Clinical Progression Free Survival | From the start of study treatment until documented progression, or death due to any cause. Assessed up to 5 years.
  Defined by a detectable post-operative prostate-specific antigen (PSA)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD FACP, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No